CLINICAL TRIAL: NCT04717726
Title: Milk Thistle and Lactobacillus Supplementation to Improve Exercise Outcomes in Obese Patients
Brief Title: Exercise, Milk Thistle, and Lactobacillus to Influence Plasma Bilirubin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyle Flack (Other)
Responsible Party: Sponsor-Investigator, Kyle Flack, Assistant professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 63147
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: Exercise; weight loss; obesity; Lactobacillus; Milk Thistle; Bilirubin
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss | interventions — milk-thistle extract; 6-phospho-beta-galactosidase; Exercise

STUDY DESIGN:
Intervention Model Description: 6 armmed, placebo controlled RCT
Who Masked: Participant, Investigator
Masking Description: Participants nor research staff working with them will know what supplement they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MT (Experimental): Participants in the MT group will be supplemented with Milk Thistle extract for 12 weeks
  Interventions: Dietary Supplement: Milk Thistle (MT)
- LAC (Experimental): Participants in the LAC group will be supplemented with Lactobacillus Gassri for 12 weeks
  Interventions: Dietary Supplement: Lactobacillus Gasseri (LAC)
- EX (Experimental): Participants in the EX group will perform aerobic exercise, 5 days per week for 12 weeks
  Interventions: Behavioral: Exercise (EX); Dietary Supplement: Control (CON)
- MT + EX (Experimental): Participants in the MT + EX group will be supplemented with Milk Thistle extract and exercise for 12 weeks
  Interventions: Dietary Supplement: Milk Thistle (MT); Behavioral: Exercise (EX)
- LAC + EX (Experimental): Participants in the LAC + EX group will be supplemented with Lactobacillus Gassri and exercise for 12 weeks
  Interventions: Dietary Supplement: Lactobacillus Gasseri (LAC); Behavioral: Exercise (EX)
- CON (Placebo Comparator): Participants in the CON group will be supplemented with maltodextrin pills made to look like the pills received by the MT and LAC groups for 12 weeks
  Interventions: Dietary Supplement: Control (CON)

INTERVENTIONS:
Dietary Supplement: Milk Thistle (MT) — Participants in the MT and EX + MT groups will be provided 900 mg of standardized milk thistle extract daily (300 mg three times per day before meals) over the 12-week regimen. We will use the standardized Jarrow Formulas Milk Thistle Veggie Caps containing 30:1 extract that is standardized to contain 80% total Milk Thistle seed flavonoids (polyphenols), including the critical Silymarin fractions isosilybinins A and B, silybinins A and B, silychristin and silydianin that is active against suppressing the UGT1A1 enzyme increasing plasma bilirubin. The capsules are free of wheat, gluten, soybeans, dairy, egg, fish/shellfish, peanuts/tree nuts, and GMOs. Rationale for using this brand: There have been inconsistencies with previous studies that did not use a standardized silymarin extract, which may have contained low levels of the active polyphenolic flavonoids in the milk thistle plant, which varies in the plant's stems, leaves, roots, and flowers.
  Arms: MT; MT + EX
Dietary Supplement: Lactobacillus Gasseri (LAC) — Participants in the LAC and LAC + EX groups will receive two doses of 3 billion CFU of lactobacillus gasseri per day for a total of 6 billion CFU, the recommended upper level for supplementation of probiotic cultures. We will use Swanson brand Lactobacillus gasseri, whose capsules are also free of wheat, gluten, soybeans, dairy, egg, fish/shellfish, peanuts/tree nuts, and GMOs. Importantly, this brand uses acid-resistant designed release capsules to improve the viability of the lactobacillus in the human stomach.
  Arms: LAC; LAC + EX
Behavioral: Exercise (EX) — Participants in the EX, EX + MT, and EX + LAC groups will complete five weekly exercise sessions on their own, expending roughly 600 kcal per session. Participants will be provided a Polar A-300 heart rate monitor programmed for their individual attributes (height, weight, age, training status, gender), which gives a real-time estimate of energy expenditure during exercise. Participants will report to the lab once per week to download the exercise sessions and verify compliance. If participants are not compliant (defined as completing 85% of their assigned exercise sessions per month), they will be disqualified. This intervention has been successfully used by Dr. Flack in multiple studies to produce significant weight loss without dietary intervention in this population with a retention rate of over 90%
  Arms: EX; LAC + EX; MT + EX
Dietary Supplement: Control (CON) — Participants in the CON and EX group will receive a placebo (maltodextrin) made to look identical to the MT and LAC capsules.
  Arms: CON; EX

SUMMARY:
The proposed clinical trial will test our hypothesis that, during exercise, red blood cell (RBC) release of heme and catabolism to bilirubin is an essential process that mediates gene responses that reduce body fat. We will evaluate whether Milk Thistle extract or Lactobacillus Gasseri extends bilirubin circulating times to decrease body fat further. Thus we will perform a 12-week, 6-armed trial with one group performing aerobic exercise 5 times per week (EX) one group receiving a Milk Thistle extract (MT), one group receiving a lactobacillus gasseri supplement (LAC), a group receiving only a placebo (CON), and groups both exercising and receiving the MT (MT + EX) and lactobacillus and exercise (LAC + EX).

DETAILED DESCRIPTION:
The investigative team's previous work has shown that BR binds to the PPARalpha protein in fat and liver tissues to activate genes that improve fatty acid oxidation via a hormone known as fibroblast growth factor-21 (FGF21). The investigators recently showed that in high capacity running rats (HCR) compared to low capacity running (LCR), in which the latter are obese, BR levels and PPARalpha-FGF21 were significantly raised in the high-capacity runners. New investigations have shown that Milk Thistle (MT) herbal supplement contains polyphenols that activate pathways that suppress the glucuronyl enzyme UGT1A1 that removes BR from the blood, improving liver function and moderately increasing BR blood levels by ~2-fold. Similar findings have been demonstrated with Lactobacillus Gasseri supplementation. Hence, there is a bilirubin-PPARalpha-FGF21 axis that can be driven by exercise and dietary supplementation. We will test whether exercise and milk thistle or exercise and lactobacillus gasseri synergistically increase bilirubin-PPARalpha-FGF21, further reducing body fat in patients with obesity.

Participants in the EX, EX + MT, and EX + LAC groups will complete five weekly exercise sessions on their own, expending roughly 600 kcal per session. Participants will be provided a Polar A-300 heart rate monitor programmed for their individual attributes (height, weight, age, training status, gender), which gives a real-time estimate of energy expenditure during exercise. Participants will report to the lab once per week to download the exercise sessions and verify compliance. If participants are not compliant (defined as completing 85% of their assigned exercise sessions per month), they will be disqualified. This intervention has been successfully used by the investigators in multiple studies to produce significant weight loss without dietary intervention in this population with a retention rate of over 90% Participants in the MT and EX + MT groups will be provided 900 mg of standardized milk thistle extract daily (300 mg three times per day before meals) over the 12-week regimen. The investigators will use the standardized Jarrow Formulas Milk Thistle Veggie Caps containing 30:1 extract that is standardized to contain 80% total Milk Thistle seed flavonoids (polyphenols), including the critical Silymarin fractions isosilybinins A and B, silybinins A and B, silychristin and silydianin that is active against suppressing the UGT1A1 enzyme increasing plasma bilirubin. The capsules are free of wheat, gluten, soybeans, dairy, egg, fish/shellfish, peanuts/tree nuts, and GMOs. Rationale for using this brand: There have been inconsistencies with previous studies that did not use a standardized silymarin extract, which may have contained low levels of the active polyphenolic flavonoids in the milk thistle plant, which varies in the plant's stems, leaves, roots, and flowers.

Participants in the LAC and LAC + EX groups will receive two doses of 3 billion CFU of lactobacillus gasseri per day for a total of 6 billion CFU, the recommended upper level for supplementation of probiotic cultures. The Swanson brand Lactobacillus gasseri will be used, as these capsules are also free of wheat, gluten, soybeans, dairy, egg, fish/shellfish, peanuts/tree nuts, and GMOs. Importantly, this brand uses acid-resistant designed release capsules to improve the viability of the lactobacillus in the human stomach.

Participants in the CON and EX group will receive a placebo (maltodextrin) made to look identical to the MT capsules.

ELIGIBILITY:
Inclusion Criteria:

* Classified as obese (BMI 30-45)
* Sedentary (do not currently exercise)
* Aged 18-50 years
* Without contraindications to exercise

Exclusion Criteria:

* Dieting for weight control
* Tobacco users
* Have a ragweed allergy
* Taking antibiotics, hypoglycemic agents, anticoagulants, statins, or NSAIDs
* Nursing, pregnant, or planning on becoming pregnant
* Supplementing with a probiotic

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Lean mass | baseline (prior to initiation of study)
  kg of lean mass will be assessed by air displacement plethysmography (BodPod, Cosmed USA)
Lean mass | 12 weeks (immediately after 12 week exercise and/or supplement intervention)
  kg of lean mass will be assessed by air displacement plethysmography (BodPod, Cosmed USA)
Fat mass | baseline (prior to initiation of study)
  kg of fat mass will be assessed by air displacement plethysmography (BodPod, Cosmed USA)
Fat mass | 12 weeks (immediately after 12 week exercise and/or supplement intervention)
  kg of fat mass will be assessed by air displacement plethysmography (BodPod, Cosmed USA)
Plasma bilirubin | baseline (prior to initiation of study)
  Plasma bilirubin will be assessed in the fasted state
Plasma bilirubin | 12 weeks (immediately after 12 week exercise and/or supplement intervention)
  Plasma bilirubin will be assessed in the fasted state
Plasma FGF21 | baseline (prior to initiation of study)
  fibroblast growth factor-21 will be assessed in the fasted state
Plasma FGF21 | 12 weeks (immediately after 12 week exercise and/or supplement intervention)
  fibroblast growth factor-21 will be assessed in the fasted state
Red blood cell count | baseline (prior to initiation of study)
  Red blood cell count will be assessed in the fasted state
Red blood cell count | 12 weeks (immediately after 12 week exercise and/or supplement intervention)
  Red blood cell count will be assessed in the fasted state
Urobilin | baseline (prior to initiation of study)
  Plasma Urobilin will be assessed in the fasted state
Urobilin | 2 weeks (immediately after 12 week exercise and/or supplement intervention)
  Plasma Urobilin will be assessed in the fasted state

SECONDARY OUTCOMES:
Liver function | baseline (prior to initiation of study)
  AST and ALT enzymes will be assessed in the fasted state to demonstrate liver health
Liver function | 12 weeks (immediately after 12 week exercise and/or supplement intervention)
  AST and ALT enzymes will be assessed in the fasted state to demonstrate liver health

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky- Nutrition Assessment Lab, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
unidentified participant data will be shared on figshare data repository
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 6 months of study completion data, for 5 years.
Access Criteria: available to public, has not been created yet